CLINICAL TRIAL: NCT02142985
Title: Respiratory Variation in Central Venous Oxygen Saturation Predicts Volume Responsiveness in Hemodynamically Unstable Patients Under Mechanical Ventilation : a Prospective Cohort Study
Acronym: VOS-HI
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, Professor, University of Monastir
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ScvO2 Flo-Trac study
Record Dates: First submitted 2014-05-06; First posted 2014-05-20 (Estimated); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Hemodynamic Instability
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- crystalloid solution (Experimental): vascular filling with 500 ml of crystalloid solution within 10 minutes
  Interventions: Drug: Sodium Chloride 0.9% Intravenous

INTERVENTIONS:
Drug: Sodium Chloride 0.9% Intravenous — vascular filling with 500 ml of crystalloid solution (sodium chloride 0.9%) over 30 minutes

SUMMARY:
Vascular filling is the main treatment of hypovolemia. Hypovolemia diagnosis can be difficult in some situations and need to be confirmed with other investigations.

Venous oxymetry based on the ScvO2 values represent a valuable way to predict responsivness to fluid filling maneuver in patients with hemodynamic instability.

DETAILED DESCRIPTION:
Vascular filling represent the milestone of the treatment of hypovolemia. Its main objective is to restore vascular volume and correct perfusion issues preventing the deleterious consequences of prolonged shock.

Hypovolemia diagnosis is easy to made in obvious clinical situations such as hemorrhagic shock, deshydratation..., but there still many diagnostic difficulties regarding latent hypovolemia especially if associated with left ventricular dysfunction.

In this situations, diagnostic of hypovolemia is hard to made and other investigations are needed.

Central venous pressure (CVP) and pulmonary occlusion artery pressure (PAPO) are the mainly used parameters for indicating vascular filling but actually many studies underline their low liability in this situation.

After vascular filling, outcome measurment is needed to evaluate the efficacity of the treatment.

Outcome measurment based on hemodynamic criteria is still insufficient. In fact, tissue hypoxia persists if the cardio - respiratory system did not adapt to the metabolic needs, that's why a pathway based on therapeutic objectives like venous oxymetry is needed.

Theorically, a filling maneuver is beneficial if associated with a ScvO2 amelioration. It reflects the amelioration of cardiac output and predicts the positive responsivness to the filling test.

ELIGIBILITY:
Inclusion Criteria:

* patients aged above 18 year old
* hemodynamic instability (hypotension or shock)

Exclusion Criteria:

* intra cardiac shunt
* severe arrythmia
* valvular regurgitation
* pacemaker
* pulmonary oedema

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
central venous oxygen saturation (ScvO2) variation | at baseline and after 10 minutes
  the ScvO2 is first measured at baseline via a central venous catheter and blood gaz, then after vascular filling (500 ml of colloid solution (Plasmagel) over thirty minutes).

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Samir, Professor, Study Director — Research Laboratory (LR12SP18) University of Monastir 5000 Tunisia
Locations (1):
- Emergency department of university hospital Fattouma Bourguiba of Monastir, Monastir, Tunisia

REFERENCES:
- [Derived] Khalil MH, Sekma A, Zhani W, Zorgati A, Ben Soltane H, Nouira S; GREAT Network. Variation in central venous oxygen saturation to assess volume responsiveness in hemodynamically unstable patients under mechanical ventilation: a prospective cohort study. Crit Care. 2021 Jul 13;25(1):245. doi: 10.1186/s13054-021-03683-6. No abstract available. PMID 34256822
- See also: official website — http://www.urgencemonastir.com